CLINICAL TRIAL: NCT06122701
Title: Cross-over Randomized Study to Determine Dose-dependent Kinetics of Thiamin in Healthy Volunteers With and Without Functional OCT1 Hepatic Transporters
Brief Title: Dose-dependent Kinetics of Thiamin in Healthy Volunteers With and Without Functional OCT1 Hepatic Transporters
Acronym: THIAMO-1
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Stefan Engeli, MD, Prof. Dr. med Stefan Engeli, University Medicine Greifswald
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IPHA-2023-007
Record Dates: First submitted 2023-11-01; First posted 2023-11-08 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Thiamin; Vitamin B1; OCT1; kinetic parameters; dose-dependency; genotypes

STUDY DESIGN:
Intervention Model Description: The study is designed as a 5-arm cross-over, open-label, randomized single oral dose comparison (5 mg, 10 mg, 50 mg, and 200 mg thiamin) and a single i.v. dose (5 mg).
Masking Description: This study is an opel-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- OCT1 deficient and wild type genotypes: 200 mg thiamin p.o. (Active Comparator): The participants are selected to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between cohort 1 and cohort 2.
  Interventions: Dietary Supplement: Thiamin p.o.
- OCT1 deficient and wild type genotypes: 50 mg thiamin p.o. (Active Comparator): The participants are selected to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between cohort 1 and cohort 2.
  Interventions: Dietary Supplement: Thiamin p.o.
- OCT1 deficient and wild type genotypes: 10 mg thiamin p.o. (Active Comparator): The participants are selected to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between cohort 1 and cohort 2.
  Interventions: Dietary Supplement: Thiamin p.o.
- OCT1 deficient and wild type genotypes: 5 mg thiamin p.o. (Active Comparator): The participants are selected to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between cohort 1 and cohort 2.
  Interventions: Dietary Supplement: Thiamin p.o.
- OCT1 deficient and wild type genotypes: 5 mg thiamin i.v. (Active Comparator): The participants are selected to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between cohort 1 and cohort 2.
  Interventions: Dietary Supplement: Thiamin i.v.

INTERVENTIONS:
Dietary Supplement: Thiamin p.o. — A single oral dose of thiamin will be administered in four intervention arms (arm 1: 200 mg, arm 2: 50 mg, arm 3: 10 mg, arm 4: 5 mg) as a drinking solution with 240 ml of still water after an overnight fast.
  A total of 15 blood samples will be taken at defined time points (baseline; 0.25; 0.5; 0.75; 1.0; 1.5; 2.0; 2.5; 3.0; 3.5; 4.0; 6.0; 8.0; 10.0; 24.0 h). At each time point, blood will be collected (4.9 ml for plasma and 2.7 ml for whole blood) to determine thiamin, TMP and TDP, and biomarkers of OCT1 transport activity. Urine will be collected during the first 10 hours after thiamin administration.
  Arms: OCT1 deficient and wild type genotypes: 10 mg thiamin p.o.; OCT1 deficient and wild type genotypes: 200 mg thiamin p.o.; OCT1 deficient and wild type genotypes: 5 mg thiamin p.o.; OCT1 deficient and wild type genotypes: 50 mg thiamin p.o.
Dietary Supplement: Thiamin i.v. — A single i.v. dose of thiamin 5 mg with 240 ml of still water after an overnight fast.
  A total of 15 blood samples will be taken at defined time points (baseline; 0.25; 0.5; 0.75; 1.0; 1.5; 2.0; 2.5; 3.0; 3.5; 4.0; 6.0; 8.0; 10.0; 24.0 h). At each time point, blood will be collected (4.9 ml for plasma and 2.7 ml for whole blood) to determine thiamin, TMP and TDP, and biomarkers of OCT1 transport activity. Urine will be collected during the first 10 hours after thiamin administration.
  Arms: OCT1 deficient and wild type genotypes: 5 mg thiamin i.v.

SUMMARY:
This study investigates the differences in thiamin (vitamin B1) kinetic parameters in two cohorts of healthy volunteers:

Cohort 1) OCT1 wild type genotypes n = 12 Cohort 2) OCT1 deficient genotypes n = 12 Participants will be selected according to their OCT1 genotypes and to achieve best matching according to sex, age, BMI, alcohol consumption, and smoking between Cohort 1 and 2, respectively.

The purpose of this study is:

1. To determine the influence of OCT1 genetic variants on dose-dependent thiamin kinetics after oral administration.
2. To elucidate whether OCT1 genetic variants impact the kinetic properties of orally vs. intravenously administered thiamin.

DETAILED DESCRIPTION:
The study is designed as a 5-arm cross-over, open-label, randomized single oral dose comparison (5 mg, 10 mg, 50 mg, and 200 mg thiamin). A fifth arm includes applying 5 mg thiamin intravenously.

A single oral dose of thiamin will be administered in four intervention arms (arm 1: 200 mg, arm 2: 50 mg, arm 3: 10 mg, arm 4: 5 mg) as a drinking solution with 240 ml of still water after an overnight fast. These four arms will be put into practice at the same time with each participant completing all four arms in random order with a wash-out period of at least one week between each arm.

After analyzing the four oral arms, we decided to administer a single i.v. dose of 5 mg thiamin in arm 5.

A total of 15 blood samples will be taken at defined time points (baseline; 0.25; 0.5; 0.75; 1.0; 1.5; 2.0; 2.5; 3.0; 3.5; 4.0; 6.0; 8.0; 10.0; 24.0 h). At each time point, blood will be collected (4.9 ml for plasma and 2.7 ml for whole blood) to determine thiamin, TMP and TDP, and biomarkers of OCT1 transport activity. At baseline, 2x 2.7 ml EDTA blood samples will be collected for DNA isolation if the particular volunteer has not had a genotypical validation in another study of our Institute.

The total amount of blood collected for each participant is 456 ml at eight kinetic visits and 10 ml at the Screening.

After intake of the thiamin solution, participants will drink 100 ml of sparkling water every hour to stimulate gastrointestinal peristalsis. After 4 hours the participants will be served a meal low in thiamin content. Urine will be collected during the first 10 hours after thiamin administration. Monitoring of blood pressure and heart rate will take place for the first 4 hours after administration. Volunteers will stay in the Clinical Research Unit of the Institute of Pharmacology for the first 10 hours after administration.

ELIGIBILITY:
Inclusion Criteria:

1. any sex
2. age between 18 and 50 years
3. OCT1 wild type: homozygous for OCT1*1 OCT "poor transporter": homozygous or heterozygous for OCT1*3, *4, *5, *6
4. understands the study purpose and design
5. contractually capable and provides signed informed consent form
6. healthy condition or mild and/or well-treated forms of allergies, asthma, hypertension, and orthopedic diseases
7. a maximum of 3 chronically taken drugs not interfering with OCT1 activity

Exclusion Criteria:

1. BMI > 32 kg/m2 and < 17 kg/m2
2. body weight < 48 kg
3. known pregnancy or lactation period
4. women: positive urine pregnancy test at screening or kinetic visit 1 of each arm
5. men: hemoglobin < 13 g/dl (8,07 mmol/l) women: hemoglobin < 12 g/dl (7,45 mmol/l)
6. elevated liver function tests (1 or more of ALAT, ASAT, yGT, Bilirubin > 2x ULN)
7. reduced renal function (eGFRMDRD < 60 ml/min/1,7 m2)
8. QTcF > 450 ms in screening ECG
9. psychiatric disease requiring recent or actual treatment
10. drug dependency at the time of visit
11. use of recreational drugs more than twice a week
12. any known hypersensitivity or allergic reactions to thiamin
13. history of severe hypersensitivity reactions and/or anaphylaxis
14. clinically proven vitamin B1 deficiency
15. individuals taking regular vitamin B1 or multi-vitamin supplements who are not willing to comply with a 48-hour washout of these supplements before each kinetic visit
16. individuals who have taken vitamin B supplements or multi-vitamins in the past 2 days before kinetic visit 1 of each arm
17. poor venous conditions that make it impossible to place a peripheral venous catheter and regularly draw blood through it

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Thiamin plasma concentrations expressed as Area under the Curve (AUC0-24 hours) | 24 hours
  Difference in thiamin plasma concentrations expressed as Area under the Curve (AUC0-24 hours) between OCT1 wild type and OCT1 deficiency cohorts (Cohort 1 vs. Cohort 2) in each dose arm

SECONDARY OUTCOMES:
Cmax of thiamin and its phosphorylated esters, TMP and TDP | 24 hours
  Differences in Cmax of thiamin and its phosphorylated esters, TMP and TDP, between the above-described cohorts in each dose arm
Tmax of thiamin and its phosphorylated esters, TMP and TDP | 24 hours
  Differences in Tmax of thiamin and its phosphorylated esters, TMP and TDP, between the above-described cohorts in each dose arm
Total and renal clearance of thiamin and its phosphorylated esters, TMP and TDP | 24 hours
  Differences in total and renal clearance of thiamin and its phosphorylated esters, TMP and TDP, between the above-described cohorts in each dose arm
Apparent volume of distribution of thiamin and its phosphorylated esters, TMP and TDP | 24 hours
  Differences in the apparent volume of distribution of thiamin and its phosphorylated esters, TMP and TDP, between the above-described cohorts in each dose arm
Plasma concentrations of known endogenous biomarkers such as isobutyrylcarnitine and propionylcarnitine | 24 hours
  Changes in plasma concentrations of known endogenous biomarkers such as isobutyrylcarnitine and propionylcarnitine measured at all time points following thiamin administration

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Engeli, Principal Investigator — Universitätsmedizin Greifswald, Institut für Pharmakologie
Locations (1):
- University Medicine Greifswald, Institute of Pharmacology, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No